CLINICAL TRIAL: NCT05962268
Title: The Effect Of Vıdeo-Based Fıstula Care Educatıon On Hemodıalysıs Patıents' Self-Care Behavıors: A Randomızed Controlled Study
Brief Title: The Effect Of Vıdeo-Based Fıstula Care Educatıon On Hemodıalysıs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Bakircay University (Other)
Responsible Party: Principal Investigator, seda şahan, Izmir Bakircay University, Izmir Bakircay University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-64577500-050.99-30751
Record Dates: First submitted 2023-06-19; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Hemolysis
Keywords: fistula care; education; self care
MeSH Terms: conditions — Hemolysis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video based education (Experimental): The video was prepared by the researchers in line with the literature. Expert opinion was obtained from 10 individuals with at least a doctorate and studies on the subject of video content. In line with expert opinions, the video content was updated and finalized. Patient education with the prepared video was provided by one of the researchers involved in the study. The video education took 20 minutes in total.
  Topics: Video recordings on of fistula care was done by the researchers in the vocational skills laboratory. The video flow plan included the introduction of the materials to be used in fistula care as well as the researcher's presentation of how to manage the fistula. Fistula care steps were performed on the simulation model. In addition, the precautions to be taken during the application and what to do in case of possible complications were also shown.
  Interventions: Other: Video based education
- Face to face education (Experimental): The patients were trained on fistula care by the researcher. Fistula care training was given to the patients in the control group using face-to-face education technique. In this training, researcher verbally explained fistula care to patients. The training was conducted one-on-one with the patient in the patient's room and lasted 10 minutes. The training was presented to the patient through the lecture method. The training was also supported by the question-and-answer method. The training was given twice, one week apart, when patients came for hemodialysis treatment after the condition of the patients on dialysis stabilized.
  Interventions: Other: Face to face education

INTERVENTIONS:
Other: Video based education — The video was prepared by the researchers in line with the literature. Expert opinion was obtained from 10 individuals with at least a doctorate and studies on the subject of video content. In line with expert opinions, the video content was updated and finalized. Patient education with the prepared video was provided by one of the researchers involved in the study. The video education took 20 minutes in total.
  Arms: Video based education
Other: Face to face education — The patients were trained on fistula care by the researcher. Fistula care training was given to the patients in the control group using face-to-face education technique. In this training, researcher verbally explained fistula care to patients. The training was conducted one-on-one with the patient in the patient's room and lasted 10 minutes. The training was presented to the patient through the lecture method. The training was also supported by the question-and-answer method. The training was given twice, one week apart, when patients came for hemodialysis treatment after the condition of the patients on dialysis stabilized.
  Arms: Face to face education

SUMMARY:
Objective: This study aimed to determine the effect of face-to-face and video-based education for fistula care on hemodialysis patients' self-care behaviors.

Methods: The study was conducted as a randomized controlled experimental study. Fistula care training was given to the patients in the control group using face-to-face education technique. Fistula care training was given to the patients in the experimental group using a video based technique.

DETAILED DESCRIPTION:
Experimental group: The researcher provided the patient education the on fistula care. In this training, the researcher first verbally explained fistula care to the patients. After the verbal training, a video recording about fistula care was shown to the patients. The patients watched the video recording during dialysis using the TV unit at the bedside. The training took 20 minutes. Patients were allowed to watch the training video twice, at a one-week interval, when they came for hemodialysis treatment after the condition of the patients on dialysis stabilized.

Topics: Video recordings on of fistula care was done by the researchers in the vocational skills laboratory. The video flow plan included the introduction of the materials to be used in fistula care as well as the researcher's presentation of how to manage the fistula. Fistula care steps were performed on the simulation model. In addition, the precautions to be taken during the application and what to do in case of possible complications were also shown.

Literature review, research results, clinicians' opinions, and experts and practices were used in editing the content of verbal training and video recording,

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or older,
* Receiving hemodialysis treatment for more than 6 months,
* Having arteriovenous fistula,
* Being able to read, understand and speak Turkish,
* Not having any physical, mental or mental disability restricting daily activities,
* Having no visual-hearing impairment, perception and psychiatric problems,
* Volunteering to participate in the study

Exclusion Criteria:

* Not having arteriovenous fistula,
* Declining to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Patient Information Form | 10 minutes
  The form consists of 12 items related to patients' gender, age, marital status, educational status, occupation, income status, duration of chronic renal failure (CRF), duration of hemodialysis, number of weekly hemodialysis, first AVF cannulation, number of AVFs, previous AVF care, and status or receiving education on kidney failure. It consists of 12 questions that determine the educational status.
Scale of Assessment of Self-Care Behaviors with Arteriovenous Fistula in Hemodialysis (ASBHD-AVF) | 10 minutes
  The scale developed by Sousa et al. (2015) can be used for the education and follow-up of patients, in addition to evaluating the care behaviors of patients towards their AVF. Each item is scored according to the its reverse statement. On the scale, a score of 1 indicates that the specified self-care behavior has never developed, and a score of 5 indicates that the specified self-care behavior is always present. The scale is concluded by summing the scores from each statement. The minimum score that can be obtained from the scale is 16, and the maximum score is 80. As the score increases, the self-care behaviors of the person improve. The validity and reliability of the scale for the Turkish population were determined by İkiz and Yıldırım Usta (2016), and the Cronbach alpha coefficient of the scale was reported to be 0.91.

CONTACTS AND LOCATIONS:
Locations (1):
- Kayseri Dialysis Center, Kayseri, Talas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Information can be obtained from the principal investigator via e-mail.